CLINICAL TRIAL: NCT04752696
Title: A Phase 2 Study of Onvansertib in Combination With Nanoliposomal Irinotecan, Leucovorin, and Fluorouracil for Second-Line Treatment of Patients With Metastatic Pancreatic Ductal Adenocarcinoma
Brief Title: Onvansertib in Combination With Nanoliposomal Irinotecan, Leucovorin, and Fluorouracil for Second-Line Treatment of Participants With Metastatic Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cardiff Oncology (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRDF-001
Record Dates: First submitted 2021-02-09; First posted 2021-02-12 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Pancreatic Ductal Adenocarcinoma
Keywords: Pancreatic Ductal Adenocarcinoma; Onvansertib; Nanoliposomal irinotecan; Leucovorin; Fluorouracil; PLK1; PLK Inhibitor
MeSH Terms: interventions — onvansertib; irinotecan sucrosofate; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Lead-in: Onvansertib + nal-IRI + leucovorin + 5-FU (Experimental): The first 3 participants will be administered onvansertib orally once a day at a dosing schedule of 12 mg/m^2 on Day 1 to Day 10 for two cycles, where each cycle is 2 weeks. Depending on the number of dose limiting toxicities (DLTs) experienced in the first 3 participants, additional participants may receive different dosing schedules, determining the dosing schedule to be used in the treatment period. Onvansertib will be administered in combination with 70 mg/m^2 nanoliposomal irinotecan (nal-IRI), 400 mg/m^2 leucovorin and 2400 mg/m^2 fluorouracil (5-FU).
  Interventions: Drug: Onvansertib; Drug: Nanoliposomal irinotecan; Drug: Leucovorin; Drug: Fluorouracil
- Treatment Period: Onvansertib + nal-IRI + leucovorin + 5-FU (Experimental): Participants will be administered onvansertib at the dosing schedule selected based on the results of the safety lead-in, in cycles of 2 weeks. Onvansertib will be administered in combination with 70 mg/m^2 nanoliposomal irinotecan (nal-IRI), 400 mg/m^2 leucovorin and 2400 mg/m^2 fluorouracil (5-FU).
  Interventions: Drug: Onvansertib; Drug: Nanoliposomal irinotecan; Drug: Leucovorin; Drug: Fluorouracil

INTERVENTIONS:
Drug: Onvansertib — Oral capsule
  Other Names: PCM-075
Drug: Nanoliposomal irinotecan — Intravenous infusion
  Other Names: Onivyde; Nal-IRI
Drug: Leucovorin — Intravenous infusion
Drug: Fluorouracil — Intravenous infusion
  Other Names: 5-FU

SUMMARY:
The main objective of this trial is to assess the efficacy of onvansertib in combination with nanoliposomal irinotecan (nal-IRI), leucovorin, and fluorouracil (5-FU) for treatment of participants with histologically confirmed metastatic pancreatic ductal adenocarcinoma (PDAC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic PDAC
* Has received 1 prior gemcitabine-based chemotherapy as first line therapy for metastatic disease. Progression after completion of neoadjuvant or adjuvant therapy of < 6 months in duration is considered 1 line of therapy for metastatic disease
* Has measurable disease according to Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1), defined as at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded) as > 20 mm with conventional techniques or as > 10 mm with spiral computed tomography (CT) scan
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1
* Must be willing and able to undergo a tissue biopsy at screening; participants who, in the opinion of the investigator, do not have tissue that is accessible for biopsy are excepted from this criterion
* Women of childbearing potential: (defined as not post-menopausal for 12 months or no previous surgical sterilization) and fertile men must agree to use adequate contraception for the duration of study participation and for 4 months after the last dose of nal-IRI. Male subjects must agree to refrain from sperm donation during the study and for 4 months after the last dose of nal-IRI
* Ability to understand and the willingness to sign a written informed consent document. Signed informed consent form must be obtained prior to initiation of study evaluations and/or activities
* International Normalized Ratio (INR) < 1.5 unless on warfarin
* Participants with prior malignancy and who were treated with no evidence of active disease more than 2 years from initial diagnosis are eligible
* Age ≥ 18 years
* Participants must have adequate organ and bone marrow function

Exclusion Criteria:

* Prior treatment with irinotecan, nal-IRI, or investigational PLK1 inhibitor
* Uncontrolled intercurrent illness including symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, and myocardial infarction within 3 months of initiation of therapy
* History of interstitial pneumonitis or interstitial lung disease
* Participants with microsatellite instability-high (MSI-H) tumors with no prior immune checkpoint inhibitor exposure
* Pregnancy or lactation
* Participant has active and uncontrolled bacterial, viral, or fungal infection(s) requiring systemic therapy
* QT interval with Fridericia's correction (QTcF) > 470 milliseconds. The QTcF should be calculated as the arithmetic mean of the QTcF on triplicate electrocardiograms (ECGs). In the case of potentially correctible causes of QT prolongation, (eg, medications, hypokalemia), the triplicate ECG may be repeated once during Screening and that result may be used to determine eligibility
* Planned concomitant use of medications known to prolong the QT/QTc interval
* Participant has undergone major surgical resection within 4 weeks prior to enrollment
* Participant received radiotherapy, surgery, chemotherapy, or an investigational therapy within 2 weeks prior to study entry
* Participant has serious medical risk factors involving any of the major organ systems such that the investigator considers it unsafe for the participant to receive an experimental research drugs
* Serious psychiatric or medical conditions that could interfere with treatment
* Major bleeding in the last 4 weeks
* More than 1 prior chemotherapy regimen administered in the metastatic setting
* Unable or unwilling to swallow oral medication
* Use of strong CYP3A4 or UGT1A1 inhibitors or strong CYP3A4 inducers. Participants currently receiving these agents who are able to switch to alternate therapy are not excluded. Inhibitors should be stopped at least one week prior to the first dose of protocol therapy and inducers should be stopped at least two weeks prior to initiation of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-12-24 (Actual); Study Completion 2024-12-24 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years

SECONDARY OUTCOMES:
Number of Participants Who Experience a Treatment-emergent Adverse Event (TEAE) | Up to 2 years
Duration of Response (DOR) | Up to 2 years
Overall Response Rate (ORR) in Participants Who Receive At Least 2 Treatment Cycles | Up to 2 years
  Each cycle is 2 weeks.
Overall Survival (OS) | Up to 2 years
Disease Control Rate (DCR) | Up to 2 years
Reduction from Baseline in Serum CA19-9 Response | Baseline up to 2 years

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Mayo Clinic Phoenix, Phoenix, Arizona
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of Kansas Medical Center, Westwood, Kansas
  - Mayo Clinic Rochester, Rochester, Minnesota
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Inova Schar Cancer Institute, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No